CLINICAL TRIAL: NCT06195579
Title: The Nurtured Heart Parenting Intervention for Children's Behavioural Problems: A Single Case Design
Brief Title: Nurtured Heart Parenting Intervention for Child Behavioural Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lincoln (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22004
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Results first posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-02

CONDITIONS: Parent-Child Relations; Child Behavior Problem
Keywords: child behavioural problems; parent training; Nurtured Heart Approach; guided self-help; single case design

STUDY DESIGN:
Intervention Model Description: Single case design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Participants receiving the intervention whilst on a waiting list for treatment as usual
  Interventions: Behavioral: Transforming the Intense Child Workbook (Glasser, 2016)

INTERVENTIONS:
Behavioral: Transforming the Intense Child Workbook (Glasser, 2016) — The NHA was delivered in a guided self-help format, using the Transforming the Intense Child workbook (Glasser, 2016) and weekly phone calls.

SUMMARY:
Behavioural problems are prevalent in children, yet the consequences can be significant for the child, family and wider society. Effective intervention is paramount in reducing the impact of childhood behavioural problems. The Nurtured Heart Approach (NHA; Glasser & Easley, 2016) is an atheoretical parenting intervention which aims to reduce childhood behavioural problems. Although used in clinical practice, there is little empirical research on the effectiveness of the NHA. The aims of the study were to examine whether the NHA reduced parent-reported child behavioural problems, reduced negative parenting practices, and increased parental reflective functioning.

The study used a multiple baseline single case design. Parents of children with behavioural problems were recruited from CAMHS waiting lists. The NHA was delivered in a guided self-help format, using the Transforming the Intense Child workbook (Glasser, 2016) and weekly phone calls. Data collection involved psychometric measures of parent-reported child behavioural problems, parenting practices and parental reflecting functioning. Measures were repeated throughout baseline and intervention phases. A follow-up four weeks after the intervention included final measure administration and a change interview. The data were graphed and visually analysed. Supplementary analysis included reliable and clinically significant change, Tau-U and percentage exceeding the median. Framework analysis was used to analyse the change interview.

ELIGIBILITY:
Inclusion Criteria:

Participants will be parents/carers of children who have been referred to National Health Service (NHS) children's services for behavioural problems. Participants will be recruited from waiting lists of NHS children's services at the two research sites in the East Midlands.

Inclusion criteria:

* The referred child is aged between three and eleven years old.
* The referred child is on a waiting list for an NHS children's service at the two research sites.
* The referred child's behavioural problems are one of the primary reasons for referral to the NHS service.
* The parent/carer identifies the referred child's behaviour as problematic.

Exclusion Criteria:

* The referred child has a diagnosis of developmental delay or learning disability.
* The family is current receiving active multi-agency involvement (e.g. social care, police or youth offending in addition to NHS services).
* The parent/carer is aged under 18.
* The parent/carer is unable to read or speak English fluently.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nima Moghaddam, Principal Investigator — University of Lincoln
Locations (1):
- University of Lincoln, Lincoln, Lincolnshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Arm
Number analyzed (Participants) | 5
Age, Customized [Number; unit: participants] — Participants were parents but the variable of interst was the age of the child referred for behavioural problems so it is the age of the referred child which is captured here.
  participants
    Age of referred child - 8 years | 1
    Age of referred child - 9 years | 1
    Age of referred child - 10 years | 1
    Age of referred child - 11 years | 2
Sex/Gender, Customized [Number; unit: participants] — Participants were parents but the variable of interst was the sex of the child referred for behavioural problems so it is the sex of the referred child which is captured here.
  participants
    Sex of referred child - male | 1
    Sex of referred child - female | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Parent-reported Child Behavioural Problems
Description: Results state the number of children for whom parents reported an improvement in behaviour using the Brief Problem Monitor (Achenbach et al., 2011).
Time Frame: Measure across the baseline phase (3 weeks), intervention phase (6 weeks) and follow up (one month post intervention)
Measure: Number; unit: participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 5
participants | 1

2. Primary Outcome: Idiographic Measure of Parent-perceived Problems
Description: Results state the number of children for whom parents reported an improvement on the ideographic goals set by parents. Measured using the PSYCHLOPS (Ainsworth et al., 2009)
Time Frame: Measured at the beginning of the baseline and follow up (one month post intervention)
Measure: Number; unit: participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 5
participants | 3

3. Secondary Outcome: Negative Parenting Practices
Description: Parents whose negative parenting practices reduced, measured using the Multidimensional Assessment of Parenting Scale (Parent and Forehand, 2017)
Time Frame: Measure across the baseline phase (3 weeks), intervention phase (6 weeks) and follow up (one month post intervention)
Measure: Number; unit: participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 5
participants | 1

4. Secondary Outcome: Parental Reflective Functioning
Description: Parents whose parental reflective function improved due to the intervention, measured using the Parental Reflective Functioning Questionnaire (Luyten et al., 2017)
Time Frame: Measure across the baseline phase (3 weeks), intervention phase (6 weeks) and follow up (one month post intervention)
Measure: Number; unit: participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 5
participants | 3

5. Secondary Outcome: Parental Wellbeing
Description: Number of parents whose wellbeing improved when measured using the SWEMWBS (Tennanet et al., 2007).
Time Frame: Measured at the beginning of the baseline and follow up (one month post intervention)
Measure: Number; unit: participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 5
participants | 2

ADVERSE EVENTS:
Time Frame: The data collection preiod - 4 months
Arm/Group | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
The study included no observational element, meaning there is no measure of the extent to which parents were using the NHA in interactions with their children. The study also highlights the limitations of measures used for the variables of interest e.g. the BPM has limited items related to externalizing behaviour but alternative measures were not appropriate for a single case design. The limitations of the measures require the results to be interpreted in the context of these shortcomings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT06195579/Prot_SAP_000.pdf